CLINICAL TRIAL: NCT06527235
Title: Efficacy of Ultrasound-monitored Meniscal Wall Betamethasone Infiltration on Pain in Relation to Degenerative Meniscal Injury: a Randomized, Double-blind, Placebo-controlled Multicenter Trial.
Brief Title: Meniscal INfiltration of Corticosteroid Guided With Ultra Sonography
Acronym: MINUS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC31/23/0387; 2023-510079-74-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Meniscus Lesion
Keywords: Betamethasone Injections; Meniscus; Ultrasonography; Randomized controlled Trial

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized vs placebo, controlled, comparative, superiority, with 2 parallel groups compared (ultrasound-guided betamethasone infiltration vs. physiological serum (identical volume) of the meniscal wall).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This trial will be double-blind (patient and evaluator). Only the physician performing the infiltration will know the status of the group assigned to the patient (experimental or placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound-guided betamethasone infiltration of the meniscal wall (Experimental): patients allocated to the experimental group will receive a single betamethasone infiltration (1mL) of the meniscal wall under ultrasound guidance.
  Interventions: Drug: ultrasound-guided betamethasone infiltration of the meniscal wall
- ultrasound-guided physiological serum infiltration of the meniscal wall (Placebo Comparator): patients allocated to the control group will receive a single placebo infiltration of isotonic saline (1mL) of the meniscal wall under ultrasound guidance.
  Interventions: Drug: ultrasound-guided isotonic saline (placebo) infiltration of the meniscal wall

INTERVENTIONS:
Drug: ultrasound-guided betamethasone infiltration of the meniscal wall — The perimeniscal injections will be guided by ultrasound with an 18 megahertz (MHz) linear probe under strict aseptic conditions. Doppler will be systematically used before the injection to identify the medial or lateral inferior geniculate artery. The first step will consist of local anesthesia with 2 ml of lidocaine injected into the subcutaneous tissues and close to the meniscus wall using a 25-gauge needle. Using an in-plane approach, a 21-gauge needle will be positioned under ultrasound guidance in the medial or lateral wall of the meniscus. Once the needle touches the meniscus wall, it will be withdrawn 1 mm, and a 1-ml injection of betamethasone into the meniscus wall will be performed.
  Arms: ultrasound-guided betamethasone infiltration of the meniscal wall
Drug: ultrasound-guided isotonic saline (placebo) infiltration of the meniscal wall — The perimeniscal injections will be guided by ultrasound with an 18 MHz linear probe under strict aseptic conditions. Doppler will be systematically used before the injection to identify the medial or lateral inferior geniculate artery. The first step will consist of local anesthesia with 2 ml of isotonic saline injected into the subcutaneous tissues and close to the meniscus wall using a 25-gauge needle. Using an in-plane approach, a 21-gauge needle will be positioned under ultrasound guidance in the medial or lateral wall of the meniscus. Once the needle touches the meniscus wall, it will be withdrawn 1 mm, and a 1-ml injection of betamethasone into the meniscus wall will be performed.
  Arms: ultrasound-guided physiological serum infiltration of the meniscal wall

SUMMARY:
The value of corticosteroid infiltration of the meniscus wall in the therapeutic strategy is not clearly defined: the data in the literature on the effectiveness of corticosteroid infiltration are heterogeneous and of low level of proof. We hypothesize that corticosteroid infiltration of the meniscal wall under ultrasound control would be effective for rapid relief of degenerative meniscal pain.

The main objective is to evaluate the efficacy of ultrasound-guided meniscal wall infiltration of betamethasone versus ultrasound-guided meniscal wall infiltration of placebo, at 1 month, on meniscal pain in the treatment of meniscal pain of degenerative origin in adult.

DETAILED DESCRIPTION:
"Meniscal pain" is a very frequent cause of consultation in orthopedics, rheumatology or sports medicine. The management of degenerative meniscal lesions has been the subject of a consensus conference by the French Authority (2008) and a recommendation by the European Society of Sports Traumatology, Knee Surgery and Arthroscopy (ESSKA 2017), which propose symptomatic medical treatment before any surgical management. Conservative medical treatment is the first-line treatment for most patients with symptomatic meniscal injuries with a wide range of therapies including rehabilitation, oral nonsteroidal anti-inflammatory drugs, joint injections of corticosteroid, hyaluronic acid, or platelet concentrates, as well as injection of corticosteroids into the posterior meniscal wall. In the therapeutic arsenal, corticosteroid infiltrations of the posterior meniscus wall are those that have been the subject of the most clinical studies, yet the data in the literature on the efficacy of these corticosteroid infiltrations are of low level of evidence. This is why the European Society of Musculoskeletal Radiology's Delphi-based consensus group on musculoskeletal imaging (ESSR) is encouraging the development of clinical research in this field with a placebo control group, in order to allow an objective validation of perimeniscal corticosteroid injection procedures in the treatment of meniscal pain of degenerative origin.

The present study is a multicenter randomized controlled trial in double blind (patient and evaluator) versus placebo. Only the physician performing the infiltration will know the status of the group assigned to the patient (experimental or placebo).

Enrollment will be prospective from the active line of patients followed in the investigating centers. A telephone pre-inclusion visit will be done at least 7 days before the inclusion visit. The inclusion visit, randomization (stratified on the centre) and infiltration will be performed on the same day. The follow-up will include a consultation at 1 month and two phone call at 7 days and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Localized knee pain with tenderness over the medial or lateral joint space reproduced on clinical examination
* Pain assessed with a VAS score > 4/10 despite first-line medical treatment including the use of tier I or II analgesics or NSAIDs.
* An MRI of the knee performed in the 6 months preceding the operation as part of the pre-treatment assessment
* Medial or lateral degenerative meniscal lesion on MRI consistent with pain, confirmed by an investigating physician
* Affiliation to the Social Security
* Free and informed consent signed by the patient

Exclusion Criteria:

* Patient under curatorship, guardianship or safeguard of justice
* Inability to speak, read or write French fluently
* Patient deprived of liberty
* Patients with psychiatric pathology
* Patient who has had an MRI showing an unstable meniscal lesion: complete vertical tear of more than 10 mm in length, capsulomeniscal disinsertion of more than 10 mm in length, complex tear, T2 hypersignal tear of liquid type with passage of liquid testifying to the spreading of the edges, tear with displaced meniscal fragment, lesion of a posterior meniscal brake, lesion of the meniscotibial or meniscofemoral attachment
* Patient with an MRI showing recent ligament injury(ies) (cruciate ligaments and/or collateral ligaments)
* History of knee trauma less than 3 months
* History of arthroscopy or open surgery of the involved knee,
* History of corticosteroid injection in the knee concerned in the 3 months preceding inclusion,
* Use of NSAIDs and oral corticosteroids during the 48 hours preceding inclusion
* Use of tier 3 analgesics for gonalgia in the 3 months prior to inclusion
* Episodes of knee instability or true locking
* Radiographic gonarthrosis with a Kellgren Lawrence stage >1 authenticated on radiographic images taken within the last 6 months.
* Known inflammatory rheumatism
* Fibromyalgia as determined by the clinical investigator
* Pregnancy and breastfeeding in progress
* Contraindication to the use of injectable corticosteroids: septic arthritis, skin lesions at the injection site, severe coagulation disorders, hypersensitivity to one of the excipients
* Contraindication to the use of systemic corticosteroids: acute infection, untreated and uncontrolled chronic infection, psychiatric or ophthalmological pathologies, unbalanced diabetes, uncontrolled hypertension
* Contraindication to the use of lidocaine: known hypersensitivity to lidocaine hydrochloride, to local anaesthetics with an amide bond or to one of the excipients, patients with recurrent porphyrias
* Patients on anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
meniscal pain at 1-month follow-up visit | month 1
  meniscal pain measured using the Visual Analog Scale (VAS) rated from 0 to 10 at 1-month follow-up visit compared to baseline VAS score

SECONDARY OUTCOMES:
meniscal pain at 3-month follow-up visit | month 3
  meniscal pain measured using the Visual Analog Scale (VAS) rated from 0 to 10 at 3-month follow-up visit compared to baseline VAS score
algo-functional scale measured by KOOS score (KNEE INJURY AND OSTEOARTHRITIS OUTCOME SCORE) at the 1-month follow-up visit | month 1
  KOOS score (algo-functional scale) at 1-month follow-up visit compared to baseline KOOS score
algo-functional scale measured by KOOS score (KNEE INJURY AND OSTEOARTHRITIS OUTCOME SCORE) at the 3-month follow-up visit | month 3
  KOOS score (algo-functional scale) at 3-month follow-up visit compared to baseline KOOS score
adverse events | month 3
  the occurrence of adverse events (AEs) and serious AEs (SAEs) up to 3 months of follow-up
Analgesic response at the 1-month follow-up visit | month 1
  Analgesic response is defined as a at least 50% reduction in pain (measured using the VAS scale) between the initial visit and the 1-month follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Marie FARUCH, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No